CLINICAL TRIAL: NCT06977763
Title: A Multicenter, Randomized, Double-blind, Positive Controlled Clinical Study on the Efficacy and Safety of Succinylated Gelatin Injection for Acute Isovolumetric Hemodilution (ANH) in Elective Surgery
Brief Title: Clinical Study on the Effectiveness and Safety of Succinylated Gelatin Injection
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Chia-tai Tianqing Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HPXMJ-III01
Record Dates: First submitted 2025-05-11; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Acute Normovolemic Hemodilution
MeSH Terms: interventions — succinylated gelatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental)
  Interventions: Drug: succinylated gelatin injection 1
- control group (Active Comparator)
  Interventions: Drug: succinylated gelatin injection

INTERVENTIONS:
Drug: succinylated gelatin injection 1 — Nanjing Chia-Tai Tianqing Pharmaceutical Company
  Arms: experimental group
Drug: succinylated gelatin injection — Gelofusine
  Arms: control group

SUMMARY:
The succinylated gelatin injection (specification: 500 mL: 20 g) developed and produced by Nanjing Chia-tai Tianqing Pharmaceutical.. is used as the experimental drug, and the succinylated gelatin injection (trade name: Gelofusine) produced by B. Braun Melsungen AG is licensed ®； Specification: 500 mL: 20 g) is used as a control drug to evaluate the clinical equivalence of two formulations in patients planning elective surgery by comparing the changes in stroke volume (SV) between 5 minutes after completion of ANH and immediately before the start of ANH.

ELIGIBILITY:
Inclusion Criteria:

1. Age range is 18 to 65 years old (including boundary values), with no gender restrictions.
2. Weight not less than 50 kg, weight not more than 100 kg, body mass index [BMI=weight (kg)/height 2 (m2)] within the range of 19.0~30.0 kg/m2 (including critical values).
3. Planned elective surgery with an estimated duration of less than 6 hours.
4. The expected ANH blood collection volume is 10% to 15% of the total blood volume.
5. Prior to enrollment, the Hb level of the subjects was ≥ 110 g/L.
6. The American Society of Anesthesiologists (ASA) has a rating of I-III.
7. Voluntarily participate in this experiment and sign a written informed consent form.

Exclusion Criteria:

1. Individuals with a history of severe cerebrovascular disease or severe mental illness, who have been deemed unsuitable by the researchers to participate in this trial.
2. Individuals who have a history of heart valve disease, aortic stenosis, and severe peripheral vascular disease (such as arteriosclerosis) and are deemed unsuitable to participate in this trial by the researchers.
3. Suffering from severe heart disease, including but not limited to a history of unstable angina, cerebrovascular accident or transient ischemic stroke (within 6 months prior to screening), myocardial infarction (within 6 months prior to screening), congestive heart failure, severe arrhythmia with poor drug control, requiring mechanical maintenance (such as pacemakers), placement of cardiac stents or New York Heart Association (NYHA) classification ≥ III at the time of screening, abnormal results on echocardiography and/or 12 lead electrocardiogram have clinical significance.
4. Patients who have previously suffered from pheochromocytoma or had poor blood pressure control during screening (SBP ≥ 160mmHg and/or DBP ≥ 100mmHg), and the researchers have determined that they are not suitable to participate in this trial.
5. Individuals with a history of liver cirrhosis or abnormal liver function during screening and deemed unsuitable for participation in this trial by the researchers: AST or ALT>2 times the upper limit of normal values; Albumin level<35 g/L; Blood bilirubin is greater than 1.5 times the upper limit of normal value.
6. Having any of the following respiratory management risks in the past: 1) history of asthma (such as allergic asthma); 2) People with sleep apnea syndrome.
7. Previously suffered from hematological disorders such as sickle cell anemia, thalassemia, etc.
8. Patients with previous or current malignant tumors (excluding non metastatic basal cell carcinoma or squamous cell carcinoma, papillary thyroid carcinoma, and cervical cancer in situ that have been cured for ≥ 5 years and do not require follow-up).
9. There is a significant risk of bleeding or coagulation disorders, and the researcher evaluates those who are not suitable to participate in this trial, including but not limited to: a) past/current thrombosis or thromboembolic events; b) Patients who stop using antiplatelet or anticoagulant drugs (such as warfarin and clopidogrel) before surgery and have not reached a half-life of 7 days or more (whichever is shorter), except for aspirin (up to 100 mg/d) and low molecular weight heparin (routine prophylactic use before surgery); c) Having a history of gastrointestinal, intracerebral hemorrhage, or other events considered severe bleeding, such as bleeding caused by the use of nonsteroidal anti-inflammatory drugs; d) When screening, PT extension>upper limit of normal value for 3 seconds or APTT extension>upper limit of normal value for 10 seconds, and the researcher evaluates it as unsuitable for surgery; e) PLT<80 × 109/L during screening.
10. Individuals with abnormal renal function assessment during screening and deemed unsuitable for participation in this trial by the researchers: Cr or BUN>1.5 times the upper limit of normal values.
11. Individuals with excessive fluid load during screening (such as systemic edema) and deemed unsuitable for participation in this trial by the researchers.
12. There were active infections with poor control during screening, and the researchers deemed it unsuitable to participate in this trial.
13. During screening, pulmonary edema, dehydration, burns, intestinal obstruction, critical illnesses such as sepsis, multiple organ failure, respiratory distress syndrome, organ transplantation, shock, etc. are combined.
14. Individuals with water electrolyte imbalance (such as hypercalcemia, hyperkalemia, etc.) during screening and deemed clinically significant by the researchers are not suitable to participate in this trial.
15. Having undergone major surgeries or surgical incisions that have not fully healed within the first 6 months of screening: Major surgeries include but are not limited to any surgeries with significant bleeding risks, prolonged general anesthesia periods, or significant traumatic injuries.
16. Received anemia related treatment, colloidal solution, and/or blood products 14 days before surgery.
17. If corticosteroids or nonsteroidal anti-inflammatory drugs cannot be discontinued within 7 days before surgery (or within 5 half lives of the drug, whichever is shorter), or if drugs that affect the subject's blood volume cannot be discontinued within 1 day before surgery (such as mannitol, etc.).
18. Individuals who are known to be allergic to any component of the investigational drug; Known to be allergic to meat, especially red meat (mammalian meat) or internal organs; Known individuals who are allergic to lactose - α -1,3-galactose; And subjects with a history of severe allergic reactions (such as urticaria, angioedema, etc.).
19. Pregnant or lactating women, as well as male subjects (or their partners) or female subjects who have a pregnancy plan during the study period until 1 month after the last use of medication, or who are unwilling to use at least one medically recognized effective contraceptive measure (such as intrauterine devices or condoms) during the study period until 1 month after the last use of medication.
20. Individuals who have participated in any other non observational clinical trials and used the study drug or device within one month prior to the trial;
21. Other situations that the researcher deems unsuitable to participate in this experiment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes in stroke volume (SV) 5 minutes after completion of ANH compared to immediately before the start of ANH | 5 minutes after the completion of ANH compared to immediately before the start of ANH

CONTACTS AND LOCATIONS:
Overall Officials: wangning shangguan, Principal Investigator — The 2nd Affiliated Hospital of Wenzhou Medical University; ting li, Principal Investigator — The 2nd Affiliated Hospital of Wenzhou Medical University